CLINICAL TRIAL: NCT01924130
Title: Increasing Breakfast Consumption and Decreasing Childhood Obesity Among Low-income, Ethnically Diverse Youth.
Brief Title: School Breakfast Policy Initiative Study
Acronym: SBPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: The Food Trust (Unknown); The School District of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20452
Record Dates: First submitted 2013-06-28; First posted 2013-08-16 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Childhood Obesity; Hunger
MeSH Terms: conditions — Pediatric Obesity | interventions — Social Marketing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- One Healthy Breakfast Program (Experimental): Classroom feeding, nutrition education lessons, social marketing, and parent outreach.
  Interventions: Other: Classroom feeding; Behavioral: Nutrition education lessons; Behavioral: Social Marketing; Behavioral: Parent outreach
- Control (No Intervention): Only receive assessments.

INTERVENTIONS:
Other: Classroom feeding — Students are fed breakfast in the classroom at the start of the school, rather than the cafeteria before school.
  Arms: One Healthy Breakfast Program
Behavioral: Nutrition education lessons — Students receive breakfast specific nutrition education lessons.
  Arms: One Healthy Breakfast Program
Behavioral: Social Marketing — A social marketing campaign designed to promote consumption of one healthy breakfast a day. The marketing includes a healthy breakfast points-based reward program designed by the students and promotional campaigns.
  Arms: One Healthy Breakfast Program
Behavioral: Parent outreach — A variety of communication methods that engage families and offer education that meets their needs, including school breakfast menus, parent newsletters, and information tables at parent-teacher meetings.
  Arms: One Healthy Breakfast Program

SUMMARY:
The purpose of this study is to develop and evaluate the effects of a school breakfast policy initiative (SBPI) on the incidence of overweight and obesity as well as breakfast patterns (both inside and outside of school) among 4th-6th grade children. The study integrates research, education and extension to promote healthy breakfast consumption among low-income children in urban schools and will leverage ongoing SNAP-Ed and the School Breakfast Program efforts.

DETAILED DESCRIPTION:
Policy makers have promoted school breakfast participation as a tool to help prevent childhood obesity. No randomized controlled trials have examined the effects of a school breakfast feeding program on obesity. We propose to develop and evaluate a School Breakfast Policy Initiative (SBPI) that combines classroom feeding, in-school nutrition education, social marketing and parent outreach. Specifically, we will promote the benefits of a healthy breakfast at school or home and deter buying "breakfast" at corner stores where purchases are high in energy, solid fats and added sugars. This intervention will be evaluated in the "real world" of urban schools that make frequent use of the SNAP-Ed and the School Breakfast Program. The specific aims are:

1. To develop the SBPI intervention within the context of SNAP Ed and the National School Breakfast Program in the School District of Philadelphia.
2. To conduct a pilot feasibility study among 4 schools (2 intervention and 2 control) to assess feasibility and acceptability.
3. To compare participants in the intervention (n=8) and comparison schools (n=8) on the incidence of overweight and obesity. We predict that intervention schools, compared to the comparison schools, will have a significantly lower incidence rate of overweight and obesity over a 2 y period.
4. To compare participants in the intervention (n=8) and comparison schools (n=8) on eating one breakfast. We predict that intervention schools, compared to the comparison schools, will have significantly greater percentage of children eating one breakfast per day over a 2 y period.

ELIGIBILITY:
Inclusion Criteria:

* 4th-8th grade Philadelphia public school students.

Exclusion Criteria:

-

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2000 (Estimated)
Dates: Start 2012-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Body Mass Index | Pilot Study: baseline (September-October 2012), 8-9 month follow up (May 2014). Main Trial: baseline (September-December 2013), 16 month follow up (January-March 2015), 32 month follow up (April-June 2016)
  BMI is calculated using students' height and weight measurements.
Breakfast Consumption habits | Pilot Study: baseline (September-October 2012), 8-9 month follow up (May 2014). Main Trial: baseline (September-December 2013), 16 month follow up (January-March 2015), 32 month follow up (April-June 2016)
  Measured using a breakfast intake questionnaire.
Hunger | Pilot Study: baseline (September-October 2012), 8-9 month follow up (May 2014). Main Trial: baseline (September-December 2013), 16 month follow up (January-March 2015), 32 month follow up (April-June 2016)
  Measured using a hunger scale questionnaire.
School meal participation rates | Every month for 34 months (September 2013-June 2016)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer O Fisher, PhD, Principal Investigator — Temple University - Center for Obesity Research and Education
Locations (1):
- Temple University - Center for Obesity Research and Education, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Polonsky HM, Bauer KW, Fisher JO, Davey A, Sherman S, Abel ML, Hanlon A, Ruth KJ, Dale LC, Foster GD. Effect of a Breakfast in the Classroom Initiative on Obesity in Urban School-aged Children: A Cluster Randomized Clinical Trial. JAMA Pediatr. 2019 Apr 1;173(4):326-333. doi: 10.1001/jamapediatrics.2018.5531. PMID 30801612
- [Derived] Dykstra H, Davey A, Fisher JO, Polonsky H, Sherman S, Abel ML, Dale LC, Foster GD, Bauer KW. Breakfast-Skipping and Selecting Low-Nutritional-Quality Foods for Breakfast Are Common among Low-Income Urban Children, Regardless of Food Security Status. J Nutr. 2016 Mar;146(3):630-6. doi: 10.3945/jn.115.225516. Epub 2016 Feb 10. PMID 26865650
- [Derived] Lawman HG, Polonsky HM, Vander Veur SS, Abel ML, Sherman S, Bauer KW, Sanders T, Fisher JO, Bailey-Davis L, Ng J, Van Wye G, Foster GD. Breakfast patterns among low-income, ethnically-diverse 4th-6th grade children in an urban area. BMC Public Health. 2014 Jun 14;14:604. doi: 10.1186/1471-2458-14-604. PMID 24928474